CLINICAL TRIAL: NCT03749330
Title: Improving Family Meetings in the Pediatric Cardiac Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-012274; K23HL141700 (NIH)
Record Dates: First submitted 2018-11-01; First posted 2018-11-21 (Actual); Results first posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Communication; Critical Illness
Keywords: cardiac intensive care unit; pediatrics; medical communication
MeSH Terms: conditions — Communication; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHOP CICU (Other): CICU Team And Loved Ones Communicating (CICU TALC)
  Interventions: Behavioral: CICU Team And Loved Ones Communicating (CICU TALC)

INTERVENTIONS:
Behavioral: CICU Team And Loved Ones Communicating (CICU TALC) — When the necessary pre-intervention clinical encounters are completed, clinicians will go through the interprofessional team training to improve communication skills and teamwork in developing care plans and communicating with families in family meetings. The first step in the study is co-design of the intervention, so it will evolve as the study continues.

SUMMARY:
This study aims to improve communication between medical teams, patients, and families in the pediatric cardiac intensive care unit. The researchers hypothesize that both improving interprofessional teamwork when preparing for family meeting and preparing families for these meetings will improve team and family satisfaction with communication. The study will involve bringing together a group of medical professionals and parents of patients to collaboratively design an intervention. In addition, the researchers will study feasibility and acceptability of the intervention and whether it impacts family and team outcomes.

DETAILED DESCRIPTION:
Context:

A large proportion of children with advanced heart disease (AHD) die in the pediatric cardiac intensive care unit (CICU), where parents describe obtaining a realistic understanding that their child had a life-limiting disease only 2 days prior to death. Delayed or inadequate communication within teams or with families may contribute to this lack of understanding (as shown in children with other serious illnesses), while interactions with pediatric palliative care specialists (PPCS) have been shown to improve communication and understanding of prognosis. The limited number of PPCS, however, means that all clinicians in the CICU must have the skills to support parental decision-making, including giving bad news and eliciting parental goals for their child.

Objectives:

1. To develop a communication skills training (CST) program for interprofessional teams in the pediatric CICU via a co-design process.
2. To evaluate CICU clinicians' perceived feasibility and acceptability of the CST.
3. To evaluate CST impact on communication skills and team function in actual family meetings.
4. To describe and evaluate parents' communication challenges in the CICU and their satisfaction with communication.
5. To determine the parents' perceived acceptability of the parent-facing aspects of the CST program.
6. Evaluate clinician fidelity to intervention plan.

Study Design:

Prospective cohort study with pre and post assessments around an intervention.

Setting/Participants:

Clinicians at the Children's Hospital of Philadelphia (CHOP) and parents of children previously hospitalized in the ICU will be invited to participate in the co-design portion of the study to develop the team and family based intervention. A separate group of volunteer attending intensivists, cardiologists, cardiac surgeons, front line clinicians, bedside nurses, and social workers from the pediatric CICU at the Children's Hospital of Philadelphia (CHOP) will undergo the intervention and participate in observed family meetings before and after the intervention. Other clinicians who are participating in an observed family meeting will also be enrolled. Parents or legal guardians and their children in the CICU who have been there for at least 7 days and are expected to stay at least another 7 days will also be consented and enrolled.

Study Interventions and Measures:

Intervention:

The intervention includes both an interprofessional team training that will include practice in communication skills of giving bad news and building team collaboration and a family oriented intervention to prepare them for family meetings.

Measures:

The Co-design process to develop the intervention will have focus groups to evaluate the interventions' content and perceived feasibility.

The impact of the intervention on CICU clinicians' perceived usefulness and satisfaction with the training will be measured with post-intervention survey and follow-up interviews.

For the actual family meetings, assessment of the impact of the intervention on communication and team function in actual family meetings pre and post-intervention will be done by coding audio recordings with validated tools and qualitative coding of content. Collaboration will be measured using the amount of time different members of different disciplines speak, and team member perception and satisfaction with collaboration will be measured using a validated tool. Fidelity of the intervention implementation will be measured by documenting behaviors of clinicians post-intervention in meetings and in chart documentation.

Parents' experiences in family meetings and perspectives on communication with the clinical team will be measured with a pre-intervention survey measuring parental mood, affect, and satisfaction with communication or with semi-structured interview. Parental perception of the CST will be measured in post-intervention surveys and acceptability interviews.

ELIGIBILITY:
Inclusion Criteria:

Participants in Co-design:

- Clinicians including attending physicians, front line clinicians (fellows, nurse practitioners, or physician assistants), bedside nurses, and social workers working at CHOP or parents of children previously hospitalized in an ICU at CHOP.

Clinicians Participating in Intervention:

- Pediatric CICU clinicians (attending intensivists, cardiologists, cardiac surgeons, front line clinicians, bedside nurses, and social workers) at CHOP who volunteer to undergo communication skills training.

Clinicians Not Participating in Intervention:

- Clinicians who plan to participate in family meetings in the pediatric CICU that will be observed by the research team.

Parent-patient Dyads Participating in the Survey or Interview:

* Parent must be the legal decision maker of a patient who has been admitted to the CHOP CICU for at least 7 days.
* Patient has been admitted to the CICU at CHOP for ≥7 days following onset of study and the medical team believes the patient will remain in the CICU for at least 7 more days OR the patient has already been admitted to the CICU for 14 days.
* Parent/guardian ≥ 18 years old.
* Child < 18 years old at time of enrollment.
* Parent/guardian is English-speaking.
* Parent/guardian has no cognitive impairments that prevent them from being a surrogate decision maker.

Exclusion Criteria:

Participants in Co-design:

- None.

Clinicians Participating in Intervention:

- Clinicians who will not participate in CHOP's CICU chronic care meeting in the following year.

Clinicians Not Participating in Intervention:

- None.

Parent-patient Dyads Participating in the Survey or Interview:

* Parent is not the legal decision maker of a patient who has been admitted to the CHOP CICU for at least 7 days.
* The medical team does not believe the patient will remain in the CICU for at least 7 more days.
* Parent/guardian < 18 years old.
* Child is ≥ 18 years old at time of enrollment.
* Parent/guardian is not English-speaking.
* Parent/guardian has cognitive impairments that prevent them from being a surrogate decision maker.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Walter, MD, PhD, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Mercer LM, Tanabe P, Pang PS, Gisondi MA, Courtney DM, Engel KG, Donlan SM, Adams JG, Makoul G. Patient perspectives on communication with the medical team: pilot study using the Communication Assessment Tool-Team (CAT-T). Patient Educ Couns. 2008 Nov;73(2):220-3. doi: 10.1016/j.pec.2008.07.003. PMID 18703306
- [Background] Pyke-Grimm KA, Degner L, Small A, Mueller B. Preferences for participation in treatment decision making and information needs of parents of children with cancer: a pilot study. J Pediatr Oncol Nurs. 1999 Jan;16(1):13-24. doi: 10.1177/104345429901600103. PMID 9989013
- [Background] Snaith RP, Zigmond AS. The hospital anxiety and depression scale. Br Med J (Clin Res Ed). 1986 Feb 1;292(6516):344. doi: 10.1136/bmj.292.6516.344. No abstract available. PMID 3080166
- [Background] Creamer M, Bell R, Failla S. Psychometric properties of the Impact of Event Scale - Revised. Behav Res Ther. 2003 Dec;41(12):1489-96. doi: 10.1016/j.brat.2003.07.010. PMID 14705607
- [Background] Anderson LA, Dedrick RF. Development of the Trust in Physician scale: a measure to assess interpersonal trust in patient-physician relationships. Psychol Rep. 1990 Dec;67(3 Pt 2):1091-100. doi: 10.2466/pr0.1990.67.3f.1091. PMID 2084735
- [Background] Epstein D, Unger JB, Ornelas B, Chang JC, Markovitz BP, Moromisato DY, Dodek PM, Heyland DK, Gold JI. Psychometric evaluation of a modified version of the family satisfaction in the ICU survey in parents/caregivers of critically ill children*. Pediatr Crit Care Med. 2013 Oct;14(8):e350-6. doi: 10.1097/PCC.0b013e3182917705. PMID 23863815
- [Background] Back AL, Arnold RM, Baile WF, Fryer-Edwards KA, Alexander SC, Barley GE, Gooley TA, Tulsky JA. Efficacy of communication skills training for giving bad news and discussing transitions to palliative care. Arch Intern Med. 2007 Mar 12;167(5):453-60. doi: 10.1001/archinte.167.5.453. PMID 17353492
- [Background] Dechairo-Marino AE, Jordan-Marsh M, Traiger G, Saulo M. Nurse/physician collaboration: action research and the lessons learned. J Nurs Adm. 2001 May;31(5):223-32. doi: 10.1097/00005110-200105000-00002. PMID 11388158
- [Background] Baggs JG. Development of an instrument to measure collaboration and satisfaction about care decisions. J Adv Nurs. 1994 Jul;20(1):176-82. doi: 10.1046/j.1365-2648.1994.20010176.x. PMID 7930118
- [Background] Barry MJ, Fowler FJ Jr, Mulley AG Jr, Henderson JV Jr, Wennberg JE. Patient reactions to a program designed to facilitate patient participation in treatment decisions for benign prostatic hyperplasia. Med Care. 1995 Aug;33(8):771-82. doi: 10.1097/00005650-199508000-00003. PMID 7543639
- [Background] Clayton JM, Adler JL, O'Callaghan A, Martin P, Hynson J, Butow PN, Laidsaar-Powell RC, Arnold RM, Tulsky JA, Back AL. Intensive communication skills teaching for specialist training in palliative medicine: development and evaluation of an experiential workshop. J Palliat Med. 2012 May;15(5):585-91. doi: 10.1089/jpm.2011.0292. Epub 2012 Mar 20. PMID 22433021

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are many different aspects of this NIH funded study which are not a clinical trial. I have included a full participant count for the funded project although there is only a subset are in the clinical trial. The clinical trial includes 2 groups: 1) Parents of hospitalized children who were in the pre and post-intervention. 2) CICU Clinicians who participated in the intervention training. Only these groups are in the participant flow and the outcome measures.
Groups:
- Parents Participating in Clinical Trial (Single Arm): Parents of hospitalized children enrolled in the pre and post-intervention arms of the study
- Clinicians Participating in Intervention Training (Single Arm): Interprofessional clinicians participated in intervention training to deploy the intervention
- Clinicians Not Participating in Intervention Training (Not CST): Clinicians Not participating in Intervention Training (not CST) but were observed in a team or family meeting and so were enrolled in the study under the same IRB.
- Pre-intervention Parents Who Only Did Interview/Survey: Parents who were enrolled in the CICU prior to the intervention who did not participate in the intervention and only completed a one time survey or interview and therefore are not considered part of the clinical trial
- Participants in the Codesign: Clinicians and parents who participated in the codesign of the intervention but did not participate in the intervention and therefore are not part of the clinical trial
- Children Patients of the Parents Enrolled in the Study: Because we collected clinical data from the medical record of patients who were children of parents enrolled in the study, these are considered enrolled participants under the IRB protocol although they did not participate in the intervention.
Period: Overall Study
Arm/Group | Parents Participating in Clinical Trial (Single Arm) | Clinicians Participating in Intervention Training (Single Arm) | Clinicians Not Participating in Intervention Training (Not CST) | Pre-intervention Parents Who Only Did Interview/Survey | Participants in the Codesign | Children Patients of the Parents Enrolled in the Study
Started | 60 | 24 | 202 | 45 | 21 | 99
Completed | 60 | 22 | 202 | 45 | 21 | 99
Not Completed | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Clinicians left work in the CICU | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This section includes participants who were not part of the clinical trial (pre-intervention parents who were only surveyed; the codesign subjects; and children of parents who were in the study) and those who did participate in the clinical trial (intervention=CST). Parents participating in the clinical trial were a combination pre and post intervention subjects given the nature of the outcomes which were about ability to collect data or outcomes only collected for post-intervention subjects.
Groups:
- Parents Participating in Clinical Trial (CST Intervention): Parents of hospitalized child enrolled in the pre and post-intervention arms of the study
- CICU Clinicians Participating in Intervention Training (CST): Interprofessional clinicians who participated in intervention training
- Clinicians Not Participating in Intervention Training (Not CST): Clinicians who were enrolled in the study because they participated in an observed team or family meeting but did not participate in the intervention training and so there are no outcome measures collected for them.
- Pre-intervention Parents Who Participated Only in the Survey or Interview, Not the CST: Pre-intervention parents who completed a one time survey or interview and were enrolled in the study for that purpose but did not participate in the family meeting that was observed as part of the intervention and therefore we have no outcome measures collected for them related to the CST.
- Participants in Codesign: Clinicians and Parents who participated in the codesign (development) of the intervention and therefore there are no outcomes measures for them.
- Children Patients of Parents Who Participated in Study: Patients who are the children of whom participated in the study. There are no outcome measures for the patient data.
- Total: Total of all reporting groups
Arm/Group | Parents Participating in Clinical Trial (CST Intervention) | CICU Clinicians Participating in Intervention Training (CST) | Clinicians Not Participating in Intervention Training (Not CST) | Pre-intervention Parents Who Participated Only in the Survey or Interview, Not the CST | Participants in Codesign | Children Patients of Parents Who Participated in Study | Total
Number analyzed (Participants) | 60 | 24 | 202 | 45 | 21 | 99 | 451
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 99 | 99
  Between 18 and 65 years | 60 | 24 | 202 | 45 | 21 | 0 | 352
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 19 | 144 | 28 | 19 | 39 | 290
  Male | 19 | 5 | 58 | 17 | 2 | 60 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 10 | 7 | 1 | 21 | 51
  Not Hispanic or Latino | 46 | 22 | 134 | 37 | 20 | 71 | 330
  Unknown or Not Reported | 3 | 1 | 58 | 1 | 0 | 7 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 26 | 1 | 1 | 3 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 13 | 2 | 5 | 7 | 1 | 19 | 47
  White | 35 | 19 | 119 | 37 | 19 | 69 | 298
  More than one race | 7 | 0 | 3 | 0 | 0 | 2 | 12
  Unknown or Not Reported | 2 | 1 | 49 | 0 | 0 | 6 | 58
Region of Enrollment [Number; unit: participants]
  United States | 60 | 24 | 202 | 45 | 21 | 99 | 451

OUTCOME MEASURES:

1. Primary Outcome: Perceived Acceptability Comparison of CICU TALC by CICU Providers Immediately After Completion of Intervention: Satisfaction Survey
Description: Acceptability of the study will be evaluated with 1 item from the Satisfaction with and Impact of the Course survey. The item is whether the training would be recommended to colleagues scored using a 4-point Likert scale (1=strongly agree to 4=strongly disagree), therefore a lower score indicates more acceptability.
Time Frame: 5 months
Population: Only clinicians were asked this question. This question was not asked of parents because it was in reference to being trained in the intervention, which only clinicians were.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm): CICU Clinicians completed intervention training to enhance their conduct of family meetings.
- Parents Participating in the Intervention (Single Arm): Parents of hospitalized children participating in the pre and post intervention
Arm/Group | CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm) | Parents Participating in the Intervention (Single Arm)
Number analyzed (Participants) | 22 | 0
score on a scale | 1.4 (0.5) |

2. Primary Outcome: Participant Retention Rates
Description: Retention rates will be tracked over time by comparing numbers of enrolled/retained subjects to numbers of those who decline to enroll or disenroll
Time Frame: 3.5 years
Population: Parents enrolled and retained in study
Measure: Count of Participants; unit: Participants
Groups:
- Parents Participating in Clinical Trial (Single Arm): Parents and their hospitalized child enrolled in the pre and post-intervention arms of the study
- CICU Clinicians Participating in Intervention Training (Single Arm): CICU clinicians who enrolled to participate in intervention training, whether they completed training or not due to disenrollment
Arm/Group | Parents Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in Intervention Training (Single Arm)
Number analyzed (Participants) | 60 | 24
Participants | 60 | 22

3. Primary Outcome: Participant Consent Rates
Description: Consent rates will be tracked over time by comparing numbers of consenting subjects to numbers of subjects who do not consent to participate
Time Frame: 3.5 years
Population: percent of all parents screened eligible for enrollment and approached who enrolled
Measure: Count of Participants; unit: Participants
Groups:
- Parents Participating in Clinical Trial (Single Arm): Parents of hospitalized child enrolled in the pre and post-intervention arms of the study
- CICU Clinicians Participating in Intervention Training (Single Arm): CICU Clinicians who were eligible to participate in the intervention training and were approached to enroll.
Arm/Group | Parents Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in Intervention Training (Single Arm)
Number analyzed (Participants) | 63 | 25
Participants | 60 | 24

4. Primary Outcome: Rates of Missing Data From Parents and Team Subjects
Description: Percent of missing data from parent and CICU team member reported survey data will be tracked throughout the study. All participants should have had data collected, therefore denominator is number of participants and the numerator is the number of participants that we received survey data from.
Time Frame: 3.5 years
Population: parents and clinicians who were supposed to complete survey data
Measure: Count of Participants; unit: Participants
Groups:
- CICU Clinicians Participating in Intervention Training (Single Arm): CICU clinicians who enrolled in intervention training
Arm/Group | Parents Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in Intervention Training (Single Arm)
Number analyzed (Participants) | 60 | 24
Participants | 59 | 22

5. Primary Outcome: Duration of Meetings Between Teams and Families
Description: Meetings will be audio-recorded and the length of each meeting measured automatically as part of analysis with NVivo qualitative coding software
Time Frame: 3.5 years
Population: Analysis of length of meeting between team and family
Measure: Mean (Standard Deviation); unit: minutes of meeting
Units Other Than Participants: meetings
Groups:
- Parent Participating in Clinical Trial (Single Arm): Parents of their hospitalized child enrolled in the pre and post-intervention arms of the study
- CICU Clinicians Participating in the Intervention Training (Single Arm): CICU Clinicians participating in the intervention training
Arm/Group | Parent Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in the Intervention Training (Single Arm)
Number analyzed (Participants) | 58 | 24
Number analyzed (meetings) | 58 | 58
minutes of meeting | 50 (20) | 50 (20)

6. Primary Outcome: Amount of Information Provided by CICU TALC as Perceived by Parent Participants in Intervention
Description: Parent participant perception of acceptability of the amount of information included in the intervention will be assessed with the amount of information item from the Patient Ratings of Shared Decision Making Program scale. Response options range from 1-3 on a 3-point Likert scale (1=less than wanted, about right, 3=more than wanted).
Time Frame: 2 years
Population: participants who completed survey data about intervention handout. CICU clinicians were not asked this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in the Intervention Training (Single Arm)
Number analyzed (Participants) | 25 | 0
score on a scale | 2.2 (0.4) |

7. Primary Outcome: Perceived Clarity of Intervention Materials of CICU TALC by Parent Participants in Intervention
Description: Parent participant perception of clarity of intervention materials will be assessed with the clarity item from the Patient Ratings of Shared Decision Making Program scale. Response options range from 1-3 on a 3-point Likert scale (1=everything clear, most things clear, 3=some/many things unclear).
Time Frame: 2 years
Population: parents who completed survey questions post-intervention. CICU Clinicians were not asked this outcome measure as it was not relevant to them.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in the Intervention Training (Single Arm)
Number analyzed (Participants) | 25 | 0
score on a scale | 1.48 (0.57) |

8. Primary Outcome: Summary Rating of CICU TALC Intervention by Parent Participants in Intervention
Description: Overall parent participant perception of the intervention will be assessed with the summary rating of intervention item from the Patient Ratings of Shared Decision Making Program scale. Response options range from 1-5 on a 5-point Likert scale (1=very positive, generally positive, neutral, somewhat positive, 5=very negative).
Time Frame: 2 years
Population: parents who completed post-intervention survey about intervention. Clinicians were not given this measure since it was not relevant to their experience of the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- CICU Clinicians Participating in Intervention Training (Single Arm): intervention training (single arm)
Arm/Group | Parents Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in Intervention Training (Single Arm)
Number analyzed (Participants) | 25 | 0
score on a scale | 1.76 (0.76) |

9. Primary Outcome: Percent of Family Meetings Adhering to Intervention Protocol
Description: For the 30 family meetings which were intended to receive the intervention (CST) we will assess the percent of those meetings which met the threshold of adhering to the intervention protocol. The denominator is the total number of observed MEETINGS in the post-intervention phase and the numerator is the number of meeting that meet the adherence threshold.
Time Frame: 2 years
Population: 30 family meeting processes were observed to determine percent of them that met a threshold of fidelity to intervention
Measure: Number; unit: percentage of meetings with fidelity
Units Other Than Participants: meetings
Groups:
- CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm): CICU Clinicians completed intervention training to enhance their conduct of family meetings and participated in post-intervention family meetings.
- Parents Participating in Clinical Trial (Single Arm): Parents of hospitalized children who participated in the pre and post intervention clinical trial
Arm/Group | CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm) | Parents Participating in Clinical Trial (Single Arm)
Number analyzed (Participants) | 24 | 60
Number analyzed (meetings) | 30 | 30
percentage of meetings with fidelity | 93 | 93

10. Primary Outcome: Percent of Team Meetings Adhering to Intervention Schedule and Protocol: Observation of Meeting
Description: Percent of Team interactions post-intervention will be monitored to assess the adherence to the intervention schedule and protocol.
Time Frame: 2 years
Population: Percent of team meetings that strictly adhered to intervention schedule and protocol. There were no families observed in these meetings so no data is entered.
Measure: Number; unit: percentage of total family meetings
Units Other Than Participants: meetings
Groups:
- Parents Participating in Clinical Trial (Single Arm): Parents of hospitalized children who participated in the pre and post-intervention clinical trial
Arm/Group | CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm) | Parents Participating in Clinical Trial (Single Arm)
Number analyzed (Participants) | 24 | 0
Number analyzed (meetings) | 30 | 0
percentage of total family meetings | 28 |

11. Primary Outcome: Feasibility of Enrollment and Retention of Participants
Description: Were we able to enroll clinicians in the intervention portion of the study and parents in the study and to what extent were they retained throughout the duration of the study.
Time Frame: 2 years
Population: Clinicians who were enrolled in the intervention and parents who were enrolled in the pre and post-intervention clinical trial. This outcome was only measured for the subjects that participated in the CST. Therefore there is no data for all other group/arms
Measure: Count of Participants; unit: Participants
Arm/Group | Parents Participating in Clinical Trial (Single Arm) | CICU Clinicians Participating in Intervention Training (Single Arm)
Number analyzed (Participants) | 60 | 24
Participants | 60 | 22

12. Secondary Outcome: Changes in CICU Providers' Use of Explicit Statements of Empathy During Family Meetings
Description: A proportion of empathic terminator statements provided by a clinician after a parental expression of negative emotion will be calculated pre and post intervention. The denominator of the proportion will be all the expressions of negative emotion by a parent and the numerator will be the instances in which a clinician responds without a statement of empathy. Because there will be a proportion calculated for all 58 meetings, we will then calculate the median proportion pre-intervention and post-intervention with an interquartile range. Empathic terminators are not desirable and therefore a lower proportion is considered a better outcome.
Time Frame: 2 years
Population: 42 clinicians who participated in a total of 58 family meetings pre and post intervention. Parents were not analyzed for this outcome.
Measure: Median (Inter-Quartile Range); unit: proportion of empathic terminators
Units Other Than Participants: meetings
Groups:
- Parents Participating in Clinical Trial: Parents of hospitalized children who participated in pre and post-intervention clinical trial
Arm/Group | CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm) | Parents Participating in Clinical Trial
Number analyzed (Participants) | 24 | 0
Number analyzed (meetings) | 58 | 0
proportion of empathic terminators
  pre-intervention | 0.5 [0.25 to 0.75] |
  post-intervention | 0.27 [0.00 to 0.6] |

13. Secondary Outcome: Changes in CICU Team Function for Communication
Description: Team function communication will be measured by changes in the Performance Assessment for Communication and Teamwork Toolset - Novice (PACT-Novice) scores. The PACT-Novice communication item is scored on a 5-point Likert scale (1-poor, 3=average, 5-excellent). Higher scores are better. We analyzed the median (IQR) differences in pre-intervention vs. Post-intervention PACT novice item "communication" scores using wilcoxon rank sum tests.
Time Frame: 2 years
Population: analyzed the median (IQR) differences in pre-intervention vs. Post-intervention PACT novice item "communication" scores using wilcoxon rank sum tests. These scores were not assigned to parents.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: meetings
Groups:
- Parents Participating in Clinical Trial (Single Arm): Parents of hospitalized children who participated in the pre or post intervention clinical trial
Arm/Group | CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm) | Parents Participating in Clinical Trial (Single Arm)
Number analyzed (Participants) | 24 | 0
Number analyzed (meetings) | 58 | 0
score on a scale
  pre-intervention | 3 [2 to 4] |
  post-intervention | 5 [5 to 5] |
Statistical Analysis 1: Comparison: CICU Clinicians Participating in Intervention Training for Clinical Trial (Single Arm); Test type: Equivalence — test of difference between pre and post; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3.5 years
Description: This was a behavioral intervention that provided communication skills training to clinicians and additional preparatory information to families before family meetings and encourage increased clarity and empathy during family meetings. The risk to clinicians and families was expected to be nearly 0. There was no monitoring for adverse reporting for elements of the study that were not a clinical trial (codesign participants, parents who only participated in the survey, and patients)
Groups:
- Parent-Patient Dyads Participating in Clinical Trial: Parents and their hospitalized child enrolled in the pre and post-intervention arms of the study
- CICU Clinicians Participating in the Intervention: CICU clinicians who participated in the training of the intervention.
Arm/Group | Parent-Patient Dyads Participating in Clinical Trial | CICU Clinicians Participating in the Intervention
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/24
Other Adverse Events (participants affected / at risk) | 0/60 | 0/24

LIMITATIONS AND CAVEATS:
This was a pilot pre-post study that was conducted with all pre-intervention data collected prior to March 2020 and all intervention and post-intervention data collected during COVID.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2021-12-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03749330/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT03749330/SAP_001.pdf
  • Informed Consent Form: Parent consent (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT03749330/ICF_002.pdf
  • Informed Consent Form: Clinician consent (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT03749330/ICF_003.pdf